CLINICAL TRIAL: NCT05069363
Title: Whole-Body Photobiomodulation Therapy for Chronic Pain: a Feasibility Trial
Brief Title: Whole-Body Photobiomodulation and Chronic Pain Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sandwell & West Birmingham Hospitals NHS Trust (Other)
Responsible Party: Principal Investigator, Dr Bethany Fitzmaurice, Clinical Fellow in Pain Medicine, Sandwell & West Birmingham Hospitals NHS Trust
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20PAIN01
Record Dates: First submitted 2021-09-02; First posted 2021-10-06 (Actual); Last update posted 2022-06-30 (Actual); Status verified 2022-06

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Intervention Model Description: A feasibility study designed as a single centre and single-armed trial with embedded qualitative component
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Intervention Group (Experimental): All participants in this feasibility trial will receive a course of whole-body photobiomodulation therapy (18 sessions over 6 weeks)
  Interventions: Device: Whole-Body Photobiomodulation Therapy

INTERVENTIONS:
Device: Whole-Body Photobiomodulation Therapy — * All participants entering the trial will receive a course of whole-body PBM therapy
  * The NovoTHOR Whole-Body PBM therapy device consists of a hinged, clamshell design with light-emitting diodes (LEDs) arranged to emit near-infrared and visible red light therapy is delivered to the entire body at once.
  * Participants will be expected to lie horizontal in the device with the lid as closed as they are comfortable with.
  * 18 sessions is the currently recommended and widely instituted and accepted practice with the NovoTHOR device.
  * The LED equipment delivers red and near infrared light therapy to the participant
  * Session 1 = 6 minutes
  * Session 2 = 12 minutes
  * Sessions 3-18 = 20 minutes
  * Timescale: 3 treatments/week for 6 weeks
  * The dosage of LED light (also known as 'fluence') will be equivalent to 25J/cm2. The device will supply a dual wavelength of red and near-infrared light with a 50:50 ratio; 660nm and 850nm respectively

SUMMARY:
Chronic pain is a common long-term condition that can affect any area throughout the body. Individuals suffering with chronic pain often have associated fatigue, sleep and mood disturbances.

Current treatments for chronic pain include a variety of both medicine-based approaches and non-medical approaches such as exercise and psychology treatments. Patients often take a combination of medications such as antidepressants and strong medications like morphine - which are not always effective, and often associated with several troublesome side effects. Despite physical activity being a common and helpful treatment, evidence shows that patients with chronic pain can find it difficult to engage for a variety of reasons. It would be helpful to see if other non-medication based approaches will be an acceptable treatment to those suffering with chronic pain.

Photobiomodulation (PBM) therapy describes a safe, non-invasive low-energy light therapy that has been successful in treating a variety of chronic pain conditions. Cells absorb light to produce a series of reactions that culminate in pain relief, reduced inflammation, and tissue repair. Most studies examining effects of PBM have consisted of a small hand-held probe focused on specific painful areas. There are a cohort of chronic pain conditions that encompass widespread throughout the back, neck and joints, such as fibromyalgia (FM). Whole-body PBM therapy is able to treat a large area of the body in a short space of time.

The main purpose of the study is to determine feasibility, with a view to guiding a definitive Randomised Controlled Trial (RCT), in terms of: feasibility of eligibility criteria, recruitment rates, acceptability of trial device in the chronic pain population, and acceptability of outcome measures.

ELIGIBILITY:
Inclusion Criteria:

Patients eligible for the trial must comply with all of the following:

1. Currently diagnosed or receiving treatment for a widespread chronic pain condition, including but not limited to:

   1. Axial pain of any origin
   2. Polyathralgia of any origin
   3. Myofascial pain of any origin
   4. A diagnosis of chronic widespread pain or FM
2. Able to provide informed written consent
3. ≥18 years
4. Able to commit time to the trial treatment schedule of 6 weeks
5. Score as low or moderate risk on the COVID-19 risk stratification tool - applicable for the duration of the pandemic

Exclusion Criteria:

1. Pregnancy
2. Severe skin diseases (e.g. skin cancer, severe eczema, dermatitis, or psoriasis)
3. Body weight ≥136kg, as per manufacturer instructions [see Appendix 3]
4. Uncontrolled co-morbidities (e.g. uncontrolled diabetes defined as HbA1c >69mmol/mol, decompensated heart failure, major psychiatric disturbance such as acute psychosis or suicidal ideation)
5. Use of systemic corticosteroid therapy including oral prednisolone or corticosteroid injections within the preceding 6 months as recommended by the manufacturer; steroids are thought to inhibit the anti-inflammatory effect of photobiomodulation therapy
6. Known active malignancy
7. Inability to enter the NovoTHOR device or lie flat for 20 minutes (either due to physical reasons or other e.g. claustrophobia)
8. Patients speaking a language for which an interpreter cannot be sought

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-01-12 (Actual); Primary Completion 2022-09 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
To determine whether eligibility criteria is either too open/restrictive by estimating eligibility and recruitment rates | 6 months
  Expressed at percentages/proportions
To investigate acceptability of the trial device and treatment schedule - by assessing refusal rates, dropout rates, trial retention rates | 6 months
  Expressed as percentages/proportions
To explore acceptability of the trial device and treatment schedule in terms of perceptions, values and opinions | 6 months
  Participant-reported experience questionnaire (qualitative)
To explore acceptability of the trial device and treatment schedule in terms of perceptions, values and opinions | 6 months
  Audio-recorded semi-structured interviews
To assess acceptability of outcome measures | 6 months
  Participant-reported experience questionnaire
Exploratory outcomes will aim to assess potential effectiveness of whole-body PBM therapy | 6 months
  Pain: Brief Pain Inventory-Short Form
  Pain severity - 4xNRS questions (0-40) Interference - 7xNRS questions (0-70)
Exploratory outcomes will aim to assess potential effectiveness of whole-body PBM therapy | 6 months
  Pain: Widespread Pain Index/Symptom Severity Score
  WPI score 0-19, SSS 0-12. Total out of 31.
Exploratory outcomes will aim to assess potential effectiveness of whole-body PBM therapy | 6 months
  Fatigue: Fatigue Severity Scale
  9 x Likert scale questions (1-7). Final score=mean
Exploratory outcomes will aim to assess potential effectiveness of whole-body PBM therapy | 6 months
  Sleep disturbance: Jenkins Sleep Questionnaire
  4 x 0-5 questions (total score out of 20)
Exploratory outcomes will aim to assess potential effectiveness of whole-body PBM therapy | 6 months
  Patient global: Patient Global Impression of Change
  1-7
Exploratory outcomes will aim to assess potential effectiveness of whole-body PBM therapy | 6 months
  Multidimensional function: Revised Fibromyalgia Impact Questionnaire (FIQR)
  21 x NRS questions (0-100)
Exploratory outcomes will aim to assess potential effectiveness of whole-body PBM therapy | 6 months
  Anxiety and Depression: Hospital Anxiety and Depression Score
  7x Likert scale questions (0-3). Total out of 21.
Exploratory outcomes will aim to assess potential effectiveness of whole-body PBM therapy | 6 months
  Tenderness: dolorimeter to apply a set pressure of <4kg/cm2 to 18 tender points
  NRS for pain at each point (0-10). MTPS/FIS score total 0 - 180
Exploratory outcomes will aim to assess potential effectiveness of whole-body PBM therapy | 6 months
  Dyscognition: Stroop Test (to assess inhibitory control and processing speed)
  Number of correct answers in 60 seconds. No negative marking
To assess participants' perceptions of randomisation, blinding and placebo therapy in a future trial | 6 months
  Participant-reported experience questionnaire (qualitative)
To assess participants' perceptions of randomisation, blinding and placebo therapy in a future trial | 6 months
  Audio-recorded semi-structured interviews

CONTACTS AND LOCATIONS:
Locations (1):
- Sandwell and West Birmingham NHS Trust, Birmingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fitzmaurice B, Heneghan NR, Rayen A, Soundy A. Whole-body photobiomodulation therapy for chronic pain: a protocol for a feasibility trial. BMJ Open. 2022 Jun 29;12(6):e060058. doi: 10.1136/bmjopen-2021-060058. PMID 35768101